CLINICAL TRIAL: NCT06959615
Title: A Multicenter, Open Phase I/IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of JAB-23E73 in Patients With Advanced Solid Tumors Harboring KRAS Gene Alteration
Brief Title: A Phase I/IIa Study of JAB-23E73 in Patients With Advanced Solid Tumors Harboring KRAS Gene Alteration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-23E73-1001
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor
Keywords: KRAS; KRAS mutation; KRAS G12C, KRAS G12D, KRAS G12V, KRAS G12S, KRAS G12A, KRAS G12D; Pan-KRAS; NSCLC; Pancreas cancer; Colorectal cancer; KRAS-mutant tumor; Targeted Therapy; JAB-23E73
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Exploration (Experimental): Monotherapy, dose escalation
  Interventions: Drug: JAB-23E73
- Phase 2a Dose Expansion (Experimental): Monotherapy, dose expansion
  Interventions: Drug: JAB-23E73

INTERVENTIONS:
Drug: JAB-23E73 — Administered orally
  Arms: Phase 1 Dose Exploration
Drug: JAB-23E73 — Administered orally
  Arms: Phase 2a Dose Expansion

SUMMARY:
This is a multicenter, open-label, phase I/IIa to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of pan-KRAS inhibitor JAB-23E73 in patients with advanced solid tumors harboring KRAS mutations or amplification. The study consists of 2 phases: Phase 1 Dose Escalation and Phase IIa Dose Expansion.

DETAILED DESCRIPTION:
Study JAB-23E73-1001 is a global multicenter, open-label Phase 1/2a study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anticancer activity of JAB-23E73 as a single agent in adult patients with advanced solid tumors with KRAS alteration. This study consists of a Phase 1a dose-escalation, followed by Phase 1b dose-expansion (dose optimization) and Phase 2a indication expansion. After completing dose-escalation, the MTD or preliminary RP2D of JAB-23E73 will be determined. Then, two of the alternative dosages of JAB-23E73 will be selected to further evaluate the efficacy, safety and PK in patients with KRAS-alternated NSCLC or other tumors, and patients may be further selected by certain/several types of KRAS-alternations based on dose escalation data. The RP2D will be determined according to the safety, efficacy and PK data from phase 1b.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytologically proven diagnosis of a locally advanced, unresectable, and/or metastatic solid tumor cancer with evidence of KRAS gene alteration (including gene mutation and wild type amplification).
2. Able to provide an archived tumor tissue sample or fresh biopsy sample.
3. Life expectancy ≥3 months at the start of treatment.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. ≥1 measurable lesion per RECIST v1.1.
6. Adequate organ function.

Exclusion Criteria:

1. Unable to swallow oral medications or with gastrointestinal dysfunction or gastrointestinal disease that significantly alters the absorption of medication.
2. Previous treatment with rat sarcoma (RAS) targeting agents.
3. Symptomatic, untreated, or actively progressing known central nervous system (CNS) metastases.
4. Impaired cardiovascular function or clinically significant cardiac disease.
5. Mean QT interval corrected using Fridericia's formula (QTcF) >470 msec.
6. Females who are pregnant or breastfeeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of participants with dose limiting toxicities (DLT) | Up to 21 days
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase. DLTs will be defined as the occurrence of any of the toxicities as described in the protocol.
Phase 2a: Objective response rate (ORR) | Up to approximately 2 years
  ORR is defined as the proportion of patients with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) per RECIST v1.1.

SECONDARY OUTCOMES:
Phase 1/2a: Adverse events | Up to approximately 2 years
  Incidence and severity of treatment-emergent Adverse Events (TEAEs), treatment-related Adverse Events (TRAEs) and serious Adverse Events (SAEs)
Phase 1/2a: Pharmacokinetic (PK): Maximum concentration (Cmax) of JAB-23E73 | Up to approximately 2 years
  PK: Cmax of JAB-23E73
Phase 1/2a: PK: Time to Maximum Concentration (Tmax) of JAB-23E73 | Up to approximately 2 years
  PK: Tmax of JAB-23E73
Phase 1/2a: PK: Area Under the Concentration Versus Time Curve (AUC) of JAB-23E73 | Up to approximately 2 years
  PK: AUC of JAB-23E73
Phase 1: ORR | Up to approximately 2 years
  ORR is defined as the proportion of patients with a BOR of confirmed CR or confirmed PR per RECIST v1.1.
Phase 1/2a: Time to Response (TTR) | Up to approximately 2 years
  TTR is defined as the time from the date of first dose of study drug to first documentation of response as assessed by the investigator per RECIST v1.1
Phase 1/2a: Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of the first dose of study drug to the date of the first documentation of progressive disease assessed by the investigator per RECIST v1.1 or death, whichever occurs first.
Phase 1/2a: Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of patients with CR, PR, or stable disease (SD) as assessed by the investigator per RECIST v1.1
Phase 1/2a: Duration of Response (DoR) | Up to approximately 2 years
  DOR is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first as assessed by the investigator.
Phase 2a: Overall Survival (OS) | Up to approximately 2 years
  OS is defined as the time from the date of first dose of study drug until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (32):
- China (32):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - National Cancer Center/Cancer Hospital- Langfang Campus, Chinese Academy of Medical Sciences and Peking Union Medical College, Langfang, Hebei
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliate of Soochow University, Suzhou, Jiangsu
  - The First Affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - ShanXi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute&Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliate Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang